CLINICAL TRIAL: NCT05730062
Title: Influence of Oxycodone on Individuals Taking an SSRI
Acronym: OXIS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: P22.052
Record Dates: First submitted 2023-01-12; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Opioid Induced Respiratory Depression; Depressive Disorder; Anxiety Disorders
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: This is a placebo controlled (oxycodone vs placebo) crossover study in patients initiating one of the following SSRIs (Paroxetine, Sertraline, Citalopram, Escitalopram)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SSRI 1 week following initiation oxycodone (Experimental): Patients will be included day 4-10 following initiation of treatment with either Paroxetine, Sertraline, Escitalopram or Citalopram and will be administered oxycodone 10 mg IR
  Interventions: Drug: Oxycodone Hydrochloride
- SSRI 1 week following initiation placebo (Placebo Comparator): Patients will be included day 25-45 following initiation of treatment with either Paroxetine, Sertraline, Escitalopram or Citalopram and and will be administered placebo comparator
  Interventions: Drug: Placebo
- SSRI 1 month following initiation oxycodone (Experimental): Patients will be included day 25-45 following initiation of treatment with either Paroxetine, Sertraline, Escitalopram or Citalopram and and will be administered oxycodone 10 mg IR.
  Interventions: Drug: Oxycodone Hydrochloride
- SSRI 1 month following initiation placebo (Placebo Comparator): Patients will be included day 25-45 following initiation of treatment with either Paroxetine, Sertraline, Escitalopram or Citalopram and and will be administered placebo comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone Hydrochloride — Oxycodone 10 mg IR
  Other Names: oxynorm
  Arms: SSRI 1 month following initiation oxycodone; SSRI 1 week following initiation oxycodone
Drug: Placebo — placebo comparator
  Arms: SSRI 1 month following initiation placebo; SSRI 1 week following initiation placebo

SUMMARY:
This study will determine whether selective serotonin reuptake inhibitors (SSRI) exacerbate opioid induced respiratory depression in patients initiating treatment for underlying conditions such as depression or an anxiety disorder. Next to paroxetine which has been evaluated in a previous study in healthy volunteers sertraline, citalopram and escitalopram will be evaluated with regards to its influence on opioid induced respiratory depression.

DETAILED DESCRIPTION:
Primary Objective:

To determine the effect of low-dose (10 mg) oxycodone versus placebo in individuals that use paroxetine on ventilation at an extrapolated end-tidal carbon dioxide concentration of 55 mmHg at 1 week (4-10 days) of SSRI treatment.

Secondary objectives:

To determine the effect of low-dose (10 mg) oxycodone versus placebo in individuals that either use sertraline, citalopram or escitalopram on ventilation at an extrapolated end-tidal carbon dioxide concentration of 55 mmHg at 1 week (4-10 days) of SSRI treatment.

To determine the effect of low dose (10 mg) oxycodone versus placebo in individuals that either use paroxetine, sertraline, citalopram or escitalopram on ventilation at an extrapolated end-tidal carbon dioxide concentration of 55 mmHg following at 1 month (25- 45 days) following initiation of SSRI treatment.

To determine whether the effects of SSRI on opioid induced respiratory depression alter during the course of treatment.

To determine the effect of low-dose oxycodone versus placebo in individuals that use and SSRI on pupil diameter.

To determine the effect of paroxetine on the pharmacokinetics of oxycodone.

Study design:

The design of the study is double-blind, placebo-controlled and cross over.

two groups will be studied: Time 1: individuals that use an SSRI for 1 week (day 4-10 after initiation of treatment); Time 2: (the same) individuals that use an SSRI for 1 month (day 25-45 after initiation of treatment); Subjects from Time 1 may transition to time 2 (preferably).

This is a crossover study. Subjects will be randomized (placebo vs oxycodone) with at least 2days in-between study days.

Subjects will be asked to take their antidepressant on t = 0 h, and will then dose the oxycodone on t = 2 h. Primary endpoint is ventilation measured at an extrapolated end-tidal PCO2 of 55 mmHg (VE55) at t = 4 h.

Prior to any antidepressant intake (t = 0) and at 1 h intervals following drug intake, the ventilatory response to hypercapnia will be measured for 6 hours. If VE55 is below 20% of baseline a further 1 or 2 measurements will be obtained

In between respiratory measurements, pupil diameter will be measured the using a handheld pupilometer. Additionally, subjects will be queried the at 1 h intervals for sedation,lightheadedness, nausea/vomiting using 11-point Likert scale from 0 (no effect) to 10 (max. possible effect).

In all subjects, a blood sample will be draw to determine the state of the CYP 2C8/3A4/2D6 gene to determine the metabolic state of the antidepressant among the subjects and relate this as covariate to our results. Additionally, 10 venous blood samples will be drawn for pharmacokinetic oxycodon analysis by Ardena (Assen). Blood will be drawn for a venipuncture in the arm or via an access line in the cubital vein. Blood sampling will be at t = 0 (blank), t = 15 min, 30 min, t = 45 min, t = 60 min, t = 120 min, t = 180 min, t = 240 min en t = 300 min.

SSRIs: the following SSRIs are planned to be studied :

* Paroxetine, dose at least 20 mg (Primary endpoint)
* Citalopram , dose at least 20 mg
* Escilatopram, dose at least 10 mg,
* Sertraline, dose at least 50 mg

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF) and able to comply with the study requirements and restrictions listed therein;
* Male and female subjects, age 18 to 75 years, inclusive;
* Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent) must have a negative serum pregnancy test prior to enrolment and must agree to use a medically acceptable means of contraception from screening through at least 1 month after the last dose of study drug;
* Body Mass Index (BMI) 18 to 35 kg/m2, inclusive;
* Stable as defined by the Investigator, based on a medical evaluation that includes the subject's medical and surgical history, physical examination, vital signs;
* Using sertraline (minimal dose 50 mg), paroxetine minimal dose 20 mg), citalopram (minimal dose 20 mg) or escitalopram (minimal dose 10 mg).

Exclusion Criteria:

* Currently meet the criteria for diagnosis of moderate or severe substance use disorder according to the DSM-5 criteria on any substances other than caffeine, or nicotine;
* Any active medical condition, organ disease or concurrent medication or treatment that may either compromise subject safety or interfere with study endpoints;
* Consume, on average, >27 units/week of alcohol in men and >20 units/week of alcohol in women (1 unit = 1 glass (250 mL) beer, 125 mL glass of wine or 25 mL of 40% spirit);
* Currently receiving medication-assisted treatment for the treatment of opioid-use disorder;
* Require on-going prescription or over-the-counter medications that are clinically relevant CYP P450 3A4 or CYP P450 2C8 inducers or inhibitors (e.g., rifampicin, azole antifungals [e.g., ketoconazole], macrolide antibiotics [e.g., erythromycin]);
* Significant traumatic injury, major surgery, or open biopsy within the prior 4 weeks of informed consent;
* History of substance use disorder;
* History of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent;
* Measured systolic blood pressure greater than 160 or less than 95 mmHg or diastolic pressure greater than 95 mmHg at screening;
* History or presence of allergic response to study medication;
* Treatment with another investigational drug within 3 months prior to dosing or having participated in more than 4 investigational drug studies within 1 year prior to screening;
* Site staff or subjects affiliated with, or a family member of, site staff directly involved in the study.
* Current use of any opioid.
* Opioid use less than 4 weeks prior to dosing with oxycodone in the current study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Ve55 Paroxetine 1 week | two hours following ingestion of the Paroxetine either oxycodone or placebo will be administered two hours following ingestion of oxycodone/placebo the change in Ve55 from baseline Ve55 will be evaluated.
  After one week of starting Paroxetine, extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be measured, followed by oxycodone or placebo ingestion. The extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be assessed two hours after oxycodone/placebo ingestion. The change from the baseline will be determined.

SECONDARY OUTCOMES:
Ve55 Sertraline, Citalopram, Escitalopram 1 week | two hours following ingestion of the Sertraline or Citalopram or Escitalopram either oxycodone or placebo will be administered two hours following ingestion of oxycodone/placebo the change in Ve55 from baseline Ve55 will be evaluated.
  After one week of starting Sertraline or Citalopram or Escitalopram, extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be measured, followed by oxycodone or placebo ingestion. The extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be assessed two hours after oxycodone/placebo ingestion. The change from the baseline will be determined.
Ve55 Paroxetine, Sertraline, Citalopram, Escitalopram at 1 month | two hours following ingestion of the Sertraline or Citalopram or Escitalopram either oxycodone or placebo will be administered two hours following ingestion of oxycodone/placebo the change in Ve55 from baseline Ve55 will be evaluated.
  After one month of starting Paroxetine, Sertraline or Citalopram or Escitalopram, extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be measured, followed by oxycodone or placebo ingestion. The extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be assessed two hours after oxycodone/placebo ingestion. The change from the baseline will be determined.
Ve55 over course Treatment | two hours following ingestion of the Sertraline or Citalopram or Escitalopram either oxycodone or placebo will be administered two hours following ingestion of oxycodone/placebo the change in Ve55 from baseline Ve55 will be evaluated.
  After one month of starting Paroxetine, Sertraline or Citalopram or Escitalopram, extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be measured, followed by oxycodone or placebo ingestion. The extrapolated ventilation at an end-tidal carbon dioxide concentration of 55 mmHg will be assessed two hours after oxycodone/placebo ingestion. The change from the baseline will be determined and will be compared to the results from 1 week following the initiation of treatment of the mentioned SSRIs
Pupillometry | Will be determined from pupillometry at t= 0,30,60,90,120,150,180,210,240,270,300 minutes
  Pupil diameter will determined at regular intervals to determine the effect of low dose oxycodone vs placebo in patients that use an SSRIs, during all visits.
Plasma concentration oxycodone | Will be determined from blood samples drawn at t= 0,15,30,45,60,120,180,240,300 minutes
  Determine the effect of paroxetine on the pharmacokinetics of oxycodone, samples will be obtained during all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD PhD, Principal Investigator — LUMC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Florian J, van der Schrier R, Gershuny V, Davis MC, Wang C, Han X, Burkhart K, Prentice K, Shah A, Racz R, Patel V, Matta M, Ismaiel OA, Weaver J, Boughner R, Ford K, Rouse R, Stone M, Sanabria C, Dahan A, Strauss DG. Effect of Paroxetine or Quetiapine Combined With Oxycodone vs Oxycodone Alone on Ventilation During Hypercapnia: A Randomized Clinical Trial. JAMA. 2022 Oct 11;328(14):1405-1414. doi: 10.1001/jama.2022.17735. PMID 36219407
- [Background] Cohen R, Finn H, Steen SN. Effect of diazepam and meperidine, alone and in combination, on respiratory response to carbon dioxide. Anesth Analg. 1969 May-Jun;48(3):353-5. No abstract available. PMID 5815096
- [Background] Geddes DM, Rudolf M, Saunders KB. Effect of nitrazepam and flurazepam on the ventilatory response to carbon dioxide. Thorax. 1976 Oct;31(5):548-51. doi: 10.1136/thx.31.5.548. PMID 11571
- [Background] Olsson M, Annerbrink K, Bengtsson F, Hedner J, Eriksson E. Paroxetine influences respiration in rats: implications for the treatment of panic disorder. Eur Neuropsychopharmacol. 2004 Jan;14(1):29-37. doi: 10.1016/s0924-977x(03)00044-0. PMID 14659984
- [Background] van der Schrier R, Roozekrans M, Olofsen E, Aarts L, van Velzen M, de Jong M, Dahan A, Niesters M. Influence of Ethanol on Oxycodone-induced Respiratory Depression: A Dose-escalating Study in Young and Elderly Individuals. Anesthesiology. 2017 Mar;126(3):534-542. doi: 10.1097/ALN.0000000000001505. PMID 28170358
- [Background] Xu L, Krishna A, Stewart S, Shea K, Racz R, Weaver JL, Volpe DA, Pilli NR, Narayanasamy S, Florian J, Patel V, Matta MK, Stone MB, Zhu H, Davis MC, Strauss DG, Rouse R. Effects of sedative psychotropic drugs combined with oxycodone on respiratory depression in the rat. Clin Transl Sci. 2021 Nov;14(6):2208-2219. doi: 10.1111/cts.13080. Epub 2021 Jun 16. PMID 34080766
- [Background] Yunusa I, Gagne JJ, Yoshida K, Bykov K. Risk of Opioid Overdose Associated With Concomitant Use of Oxycodone and Selective Serotonin Reuptake Inhibitors. JAMA Netw Open. 2022 Feb 1;5(2):e220194. doi: 10.1001/jamanetworkopen.2022.0194. PMID 35201310